CLINICAL TRIAL: NCT02422875
Title: Comparative Autoantibody and Immunologic Cell Marker Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Ignacio Sanz, Professor, Emory University
Other Study IDs: IRB00058515; 5R37AI049660 (NIH)
Record Dates: First submitted 2015-04-17; First posted 2015-04-21 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Autoimmune Diseases; Lupus Erythematosus, Systemic; Communicable Diseases
Keywords: Sjögren's Syndrome; Scleroderma; Myositis; Juvenile Idiopathic Arthritis; Rheumatoid Arthritis; Inflammatory Arthritis; Undifferentiated Connective Tissue Disease; Idiopathic thrombocytopenic purpura; Graft vs Host Disease; Autoimmune Lymphoproliferative Syndrome; Immunoglobulin G4 (IgG4)-related disease; Hepatitis C; Epstein Barr Virus (infectious mononucleosis - EBV); Sepsis; Guillain-Barre syndrome; Mycoplasma pneumoniae; Human Immunodeficiency Virus
MeSH Terms: conditions — Autoimmune Diseases; Lupus Erythematosus, Systemic; Communicable Diseases; Sjogren's Syndrome; Scleroderma, Diffuse; Myositis; Arthritis, Juvenile; Arthritis, Rheumatoid; Arthritis; Undifferentiated Connective Tissue Diseases; Purpura, Thrombocytopenic, Idiopathic; Graft vs Host Disease; Autoimmune Lymphoproliferative Syndrome; Immunoglobulin G4-Related Disease; Hepatitis C; Epstein-Barr Virus Infections; Sepsis; Guillain-Barre Syndrome; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Biospecimen Retention: Samples With DNA — Acquisition and storage of blood and bone marrow samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Healthy Controls: Subjects are healthy persons without any autoimmune conditions or infectious diseases
- Autoimmune Disease: Subjects diagnosed with autoimmune disease including but not limited to: Systemic Lupus Erythematosus (SLE), Sjögren's Syndrome (SS), Scleroderma, Myositis, Juvenile Idiopathic Arthritis (JIA), Rheumatoid Arthritis (RA), inflammatory arthritis, undifferentiated connective tissue disease, idiopathic thrombocytopenic purpura (ITP), Graft vs Host Disease (GVHD), Autoimmune Lymphoproliferative Syndrome (ALPS) and IgG4-related disease
- Infectious Disease: Subjects diagnosed with an infectious disease including but not limited to: Hepatitis C, Epstein Barr Virus (infectious mononucleosis - EBV), Sepsis, Guillain-Barre syndrome (GBS), Mycoplasma pneumoniae or Human Immunodeficiency Virus (HIV)
- Autoimmune - Family: Subjects have a brother, sister, mother, father, or child with an autoimmune disease
- Vaccination: Subjects have received or will receive a vaccination as part of regular standard of care from their healthcare provider or other outside source

SUMMARY:
The purpose of this study is to compare immune phenotype, function, and specificity of B lymphocytes from different developmental stages in autoimmune patients to B cells from infectious disease patients and healthy controls.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is an autoimmune disease (in autoimmune illness, the immune system in the body attacks it's own cells, leading to illness). It is not completely understood how this disease develops in the body. In a normal person, there is a tolerance of antigens (substances that make antibodies, which protect the body from disease-causing agents). Research in mice suggests that defects in certain types of cells can make the body lose this tolerance, therefore recognizing antigens made in the body as foreign, and mounting an immune response to the "self", thus causing autoimmune disease. In this study, the researchers will look at these potentially defective cells in people with SLE and other autoimmune diseases and compare them to cells in healthy participants, as well as looking at the blood of first-degree relatives of people with autoimmune disease.

The study involves blood draws and bone marrow aspirates. Participants may be asked to donate 2/3 to about 9 tablespoons of blood. The volume of blood needed will depend on the experiment being done as different numbers of cells are necessary to run different experiments. Study participants may return for additional blood draws will not donate blood more than twice a week, and will not have more than 16 tablespoons of blood drawn in a one-month period. Participants donating bone marrow will have about 3 ½ tablespoons of bone marrow obtained, which will be drawn with a large needle from the bone located in the back of the hip. Bone marrow participants may be asked to donate up to 7 tablespoons of blood as well, in order to correlate the blood with the bone marrow sample and the populations of cells residing in each. Participants donating bone marrow may donate more than once, but must wait a minimum of 8 weeks between donations.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent by the subject or, if the subject is unable to provide informed consent, the subject's legal representative may provide consent.
* Subjects can be of either gender
* Subjects with autoimmune diseases, and Systemic Lupus Erythematosus (SLE) patients will fulfill the American College of Rheumatology Classification criteria for SLE to be determined by their treating physician but may have incomplete criteria (<4 items). SLE patients are not restricted by treatment or by disease activity as determined by Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) or Systemic Lupus Activity Measure (SLAM) score

  1. Subjects with acute exacerbations of their disease, including hospitalized patients
  2. First-degree relatives of subjects with active disease
* Subjects who have received or will receive a vaccination may be enrolled for bone marrow aspirates before and/or after vaccination. Vaccination will have been done by the subject's healthcare provider or through another outside source.
* Subjects may have a screening blood draw performed in cases where a certain subset of cells or antibody titer is desired. This may be followed by additional blood draws and/or bone marrow aspiration after the ideal candidates have been identified.
* Subjects who have been diagnosed with HIV or another infectious disease
* Subjects taking biologic and/or immune modulatory agents in diseases such as cancer, allergy, and pulmonary diseases will be enrolled.
* Healthy controls must be free of acute or chronic disease at the time of bone marrow donation. Healthy controls that are first-degree relatives of subjects with active disease will be enrolled as well.

Exclusion Criteria:

* Poor venous access
* Subjects who have had side effects to local anesthetics such as lidocaine and who are on blood thinners such as warfarin
* Normal controls must be free of acute or chronic diseases or medications that may affect the assay (as determined by the investigator).
* For subjects donating bone marrow, insufficient access to the iliac crest such that the periosteum and bone is hindered based on normal aspiration procedures.
* Pregnant or lactating women may not donate bone marrow.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Subjects with certain autoimmune conditions or if subjects have brothers, sisters, mother, father, or children with an autoimmune condition
  * Subjects with certain infectious diseases
  * Subjects who are without an autoimmune condition or infectious disease
  * Subjects who have received or will receive a vaccination as part of their regular standard of care from one of their healthcare providers
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2012-08; Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Distribution of autoreactive B cells within bone marrow | Baseline
  B cells will be analyzed using flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Ignatio Sanz, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Grady Health System, Atlanta, Georgia